CLINICAL TRIAL: NCT04136821
Title: The Long-term Effects of Oceanix™ Supplementation on Oxidative Stress, Performance, Body Composition and Safety Metrics
Brief Title: The Long-term Effects of Oceanix™ on Resistance Training Adaptations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Science & Performance Institute (Industry)
Collaborators: Lonza Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASPI0519
Record Dates: First submitted 2019-10-16; First posted 2019-10-23 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Oxidative Stress; Muscle Strength; Resistance Training; Body Composition; Muscle Damage
Keywords: Oxidative Stress; Muscle Strength; Resistance Training; Antioxidants
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Double-blind, parallel, randomized, placebo-controlled trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants will engage in a 6 week, whole-body, resistance training program 3-5 days per week will consuming a visually identical placebo (25mg hydroxypropyl methylcellulose) 30 minutes prior to exercise on training days or with the first meal of the day on non-training days.
  Interventions: Other: Resistance Training
- Oceanix™ (Experimental): Participants will engage in a 6 week, whole-body, resistance training program 3-5 days per week will consuming a the treatment condition (Oceanix™) 30 minutes prior to exercise on training days or with the first meal of the day on non-training days.
  Interventions: Dietary Supplement: Oceanix; Other: Resistance Training

INTERVENTIONS:
Dietary Supplement: Oceanix — Ingredient contains highly active antioxidant enzymes, including superoxide dismutase (SOD), as well as essential fatty acids, vitamins, amino acids and minerals.
  Arms: Oceanix™
Other: Resistance Training — 6 weeks of supervised and programmed whole body resistance training, performed 3-5 times per week.

SUMMARY:
This study will examine the effects of Oceanix™, an antioxidant supplement, on muscle performance, immune and endocrine function, recovery and safety in participants undergoing resistance training. Measures of muscle performance will include isometric testing in the bench-press and mid-thigh pull and ground reaction forces in the counter movement- and squat-jump. Markers of immune function will include salivary immunoglobulin A (IgA) as well as serum total antioxidant capacity (TAC) and superoxide dismutase (SOD) while endocrine function will be measured by salivary cortisol and testosterone. Recovery will be measure by plasma creatine kinase (CK) and perceptual measures will be assessed using a validated perceived recovery status (PRS) scale. Safety metrics will be indicated by a comprehensive metabolic panel (CMP), complete blood count (CBC), and urinalysis (UA). Additionally, the modified Borg Rating of Perceived Exertion (RPE) will be administered following each training session to grade physical exertion and monitor progression of the training protocol.

DETAILED DESCRIPTION:
This study will examine the effects of Oceanix™, an antioxidant supplement, on muscle performance, immune and endocrine function, recovery and safety in participants undergoing resistance training. Measures of muscle performance will include isometric testing in the bench-press and mid-thigh pull and ground reaction forces in the counter movement- and squat-jump. Markers of immune function will include salivary immunoglobulin A (IgA) as well as serum total antioxidant capacity (TAC) and superoxide dismutase (SOD) while endocrine function will be measured by salivary cortisol and testosterone. Recovery will be measure by plasma creatine kinase (CK) and perceptual measures will be assessed using a validated perceived recovery status (PRS) scale. Safety metrics will be indicated by a comprehensive metabolic panel (CMP), complete blood count (CBC), and urinalysis (UA). Additionally, the modified Borg Rating of Perceived Exertion (RPE) will be administered following each training session to grade physical exertion and monitor progression of the training protocol.

This study will be a double blind parallel, randomized placebo-controlled trial. The investigators will request participation from 25 male and female participants (40-60 % mixture of each) ranging from 18 to 45 years old who are active (i.e. 30 minutes per week of vigorous activity classified as greater than 75 % of their HR max 3 days • week-1). The exclusion criteria will include having a BMI of 30 or more kg/m²; having cardiovascular, metabolic, or endocrine disease; undergone surgery that affects digestion and absorption, smoking, drinking heavily (> 7 and > 14 drinks per week for women and men, respectively), women who are pregnant or planning to be pregnant; taking medication to control blood pressure, lipids, and blood glucose; have taken or currently taking anabolic-androgenic steroids. The investigators will also exclude individuals using antioxidant supplements, NSAIDS, or nutritional supplements known to stimulate recovery or muscle mass gains, heart disease, prescription medications, dietary supplements that enhance body strength, muscle, immune function, muscle recovery, or soreness. Additionally, individuals cannot have allergies for seaweeds or marine sources or any dietary supplements or take any psychiatric supplements or blood thinners.

Participants will be baselined and post-tested at week zero and again after 6 weeks of training, respectively. However, on weeks 2 and 5, participants will experience an overreaching phase to induce stress, and run through specific tests to gauge recovery at the end of those specific weeks. Variables collected at these time points are described below.

Primary variables:

* Muscle, fat mass, and bone density as indicated on DXA
* Upper body strength, velocity, and power on the bench press.
* Lower body strength and power on a dual force plate.
* Vertical jump performance on a dual force plate.
* Movement mechanics and stability using a combination of motion analysis and a dual force plate.

Secondary Variables

* CBC, CMP, Urinalysis
* Vital signs (blood pressure)
* Adverse Events Scale
* PRS and RPE scales

At the end of weeks 2 and 5 participants will be examined for their perceived recovery, soreness, serum markers of muscle damage (creatine kinase), and oxidative stress markers (SOD and Total Antioxidant Status). The rationale for the time points is to introduce extreme stressors in the early and late stages of the training protocol. Variables collected at these time points are described below.

Secondary variables

* Muscle damage (blood creatine kinase), soreness, and recovery.
* Immune function (IGA) , endocrine function (cortisol and testosterone), and oxidative stress (SOD and total antioxidant status).
* PRS scale

ELIGIBILITY:
Inclusion Criteria:

* Physically active males and females aged 18 to 45 years.
* Volunteers are deemed active if they engage in 30 minutes of vigorous activity, classified as greater than 75 % of their HR max, 3 days • week-1.

Exclusion Criteria:

* > BMI of 30 or more kg/m²
* Cardiovascular, metabolic, or endocrine disease
* Undergone surgery that affects digestion and absorption
* Smoking
* Drinking heavily (> 7 and > 14 drinks per week for women and men, respectively)
* Women who are pregnant or planning to be pregnant
* Taking medication to control blood pressure, lipids, and blood glucose
* Have taken or currently taking anabolic-androgenic steroids
* Individuals using antioxidant supplements, NSAIDS, or nutritional supplements known to stimulate recovery or muscle mass gains, heart disease, prescription medications, dietary supplements that enhance body strength, muscle, immune function, muscle recovery, or soreness
* Allergies for seaweeds or marine sources

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2019-11-15 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Changes in muscle strength | Pre, Week 2, Week 5, Week 6
  Assessed by isometric mid-thigh pull and isometric bench-press
Changes in muscle power | Pre, Week 2, Week 5, Week 6
  Assessed through ground reaction forces during countermovement- and squat-jumps on a force plate.
Total Antioxidant Capacity (TAC) | Pre, Week 2, Week 5, Week 6
  Experimental outcome examining total antioxidant capacity in fasted whole blood samples. The TAC measures the overall collective power of the blood to neutralize free radicals.
Superoxide Dimutase (SOD) | Pre, Week 2, Week 5, Week 6
  Experimental outcome examining superoxide dimutase in fasted whole blood samples. This is another protective antioxidant enzyme measured from whole blood.
Creatine Kinase (CK) | Pre, Week 2, Week 5, Week 6
  Experimental outcome examining creatine kinase in fasted whole blood samples. This is biomarker an indirect measure of muscle damage.
Body Composition | Pre and Week 6
  Body Composition will be assessed via dual-energy x-ray absorptiometry (DXA). Using this method, changes in total-, lean-, and fat-mass will be examined.

SECONDARY OUTCOMES:
Rating of Perceived Exertion (RPE) | Following every resistance training session throughout the study.
  Assessed through a visual analog scale (modified Borg Scale) numbered 0-10 with visual descriptors. For example, at 0 the descriptor is "rest" and at 10 the descriptor is "maximal exertion".
Perceived Recovery Status (PRS) | Prior to every resistance training session throughout the study.
  Assessed through a visual analog scale numbered 0-10 with visual descriptors. For example, at 0 the descriptor is "very poorly recovered/extremely tired" and at 10 the descriptor is "very well recovered/highly energetic".
Immunoglobulin A (IgA) | Pre, Week 2, Week 5, Week 6
  Experimental outcome examining the concentration of IgA in fasted saliva samples.
Cortisol | Pre, Week 2, Week 5, Week 6
  Experimental outcome examining the concentration of Cortisol in fasted saliva samples.
Testosterone | Pre, Week 2, Week 5, Week 6
  Experimental outcome examining the concentration of testosterone in fasted saliva samples.
Complete Blood Count | Pre and Week 6
  Complete blood count with differential will be assessed via fasted whole blood samples.
Comprehensive Metabolic Panel | Pre and Week 6
  Comprehensive metabolic panel will be assessed via fasted whole blood samples.
Urinalysis | Pre and Week 6.
  Urinalysis gross examinations will be conducted prior to and at the completion of the study (Week 6).

OTHER OUTCOMES:
Resting Systolic Blood Pressure | Pre and Week 6
  Change in resting systolic blood pressure.
Resting Diastolic Blood Pressure | Pre and Week 6
  Change in resting diastolic blood pressure.

CONTACTS AND LOCATIONS:
Locations (1):
- Applied Science & Performance Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No